CLINICAL TRIAL: NCT02047877
Title: Investigation of Airway Inflammatory Response During an Acute Respiratory Illness in Pediatric Patients With Respiratory Failure
Brief Title: Airway Inflammatory Response During Illness in Children With Respiratory Failure
Status: Withdrawn | Type: Observational
Why Stopped: Study concept vacated due to sample collection issues
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 13-2784
Record Dates: First submitted 2014-01-25; First posted 2014-01-28 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Acute Respiratory Failure; Acute Respiratory Infection; Acute Respiratory Distress Syndrome
Keywords: Respiratory Secretions; Tracheal Secretions; Bronchial Secretions; NonBronchoscopic BAL; Interleukin 10; Interleukin 12p70
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Will bank all remaining serum, tracheal secretion, and bronchial secretion de-identified for purposes of future unknown scientific studies designed at examining respiratory secretions in this defined pediatric population.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Respiratory Illness: Previously healthy patients admitted with acute respiratory illness who are then intubated requiring mechanical ventilator support. Endotracheally intubated patients of age 37 weeks gestation through 17 years with an acute respiratory illness in the absence of existing cardiopulmonary disease, tracheostomy, or immunocompromised condition. Tracheal aspirates (TA), bronchial fluid (nb-BALF), and blood are collected within 48-hours following endotracheal intubation. All three samples are collected again at two additional time points following intubation: between days 3-4 and between days 5-7, so long as the patient remains endotracheally intubated.

SUMMARY:
The purpose of this study has two major goals: 1) to measure the amount of two specific hormones interleukin (IL)-10 and interleukin (IL)-12p70 in mucous and blood; and 2) compare the hormone levels in two specific areas of the lung called the trachea (upper airway) and the bronchioles (lower airway). The hormones IL-10 and IL-12p70 are cytokines, special hormones cells use to communicate with each other during inflammation or infection. Cytokines can be measured in mucous and blood. The balance of one cytokine compared to another help doctors to understand how people respond differently to infection. Unfortunately, the amount of IL-10 and IL-12p70 is not known in children, especially children with a lung infection. In addition, we do not know if the balance of these cytokines differ in various regions of the lung. We believe the balance of IL-10 and IL-12p70 is similar whether measured in the upper or lower airways.

DETAILED DESCRIPTION:
This study is designed to measure the concentration and describe the distribution of cytokine IL-10 and IL-12p70 in a previously healthy pediatric population suffering direct lung injury by an infectious etiology, not yet described in the literature.

In addition, this study seeks to determine whether tracheal aspirates (TA) obtained in early acute respiratory failure can be substituted for distal airway aspirates, obtained by non-bronchoscopic broncho-alevolar lavage (nb-BAL), for the purposes of investigating markers of inflammation. We will compare the ratio of IL-10 to IL-12p70 at each time point measured in tracheal secretion, bronchial secretion, and blood to assess for sample equivalence.

Finally, this study will affirm the safety profile for repeated nb-BAL, establish a protocol for respiratory sample collection and storage for future larger scale studies, and generate feasibility data regarding consent rate, estimates of data completion, and fraction of missing data for us to determine whether a future study involving the ratio of IL-10 to IL-12p70 can be used as a predictor of acute respiratory distress syndrome (ARDS) in this population.

The data generated by this study regarding safety, comparison of nb-BAL and TA, and cytokine concentrations will be used as preliminary data informing the design of a larger multicenter study testing the hypothesis that IL-10 and IL-12p70 levels in airway secretions can predict risk for ARDS in this population. This may be approached via application to the Pediatric Acute Lung Injury and Sepsis (PALISI) clinical research network group.

ELIGIBILITY:
Inclusion Criteria:

* Previously healthy
* Age 37 weeks gestation through 17 years
* Presumed respiratory infection
* Intubated <48 hours

Exclusion Criteria:

* Trauma, Drowning, Pancreatitis, or Sepsis not originating from a pulmonary infection.
* Pre-existing chronic disease including:
* congenital heart disease or acquired cardiomyopathy
* pulmonary hypertension
* restrictive lung disease
* cystic fibrosis
* asthma controlled with chronically inhaled steroids
* Tracheostomy
* Immunocompromised including chronic steroid use within last month
* Oncological condition except conditions in active remission not requiring maintenance chemotherapy.
* Intubated patient with an endotracheal tube <3.5 mm
* Patients with persistent SpO2 <90% despite adequate ventilator support, or patients deemed too unstable to undergo mini-BAL by the clinical care team

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Previously healthy patients presenting to UNC with respiratory failure presumptively caused by a primary lung infection will be screened. Only those patients intubated within 48-hours of potential enrollment and between the ages of ≥37 weeks gestation and 17 years will be considered. For purposes of this study, acute respiratory illness is defined as having upper respiratory infection symptoms and/or lower respiratory tract infection. Patient should have fever (>38 oC) OR leukocytosis / leukopenia (>10,000 or <2,000) AND any of the following: tachypnea, hypoxia (saturation <97%), cough, congestion, rhinorrhea, abnormal lung exam findings, or infiltrate on chest x-ray.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Mean log transformed IL-10:IL-12p70 ratio in tracheal secretion, bronchial secretion, and serum within 48-hours of mechanical ventilation | Within 48 hours of mechanical ventilation
  Tracheal aspirates (TA), bronchial fluid (nb-BALF), and blood are collected within 48-hours following endotracheal intubation. All three samples are collected again at two additional time points following intubation: between days 3-4 and between days 5-7, so long as the patient remains endotracheally intubated. Three time points were chosen to show consistency in ratio of IL-10 to IL-12p70 between TA and nb-BALF throughout the first week of endotracheal intubation. If a patient is extubated before day 7 all sample collection will stop. No samples will be obtained after 7 days of intubation as we are focusing on the acute phase of lung injury only. An ELISA assay is performed to measure the concentration of IL-10 and IL-12p70 for ratio comparison.

SECONDARY OUTCOMES:
Blood oxygenation saturation and hemodynamic changes following non-bronchoscopic BAL | Baseline through 1-hour post procedure
  Pulse Oxygen Saturation (SpO2), heart rate (HR), blood pressure (BP), and cardiac rhythm are continuously monitored per clinical routine in intubated patients. These parameters will be recorded pre-procedure then monitored over the 1 hour post-procedure. Transient and inconsequential changes in these parameters are expected. The following changes will be considered adverse events and reported to data safety monitor (DSM):
  1. Persistent (>10 minute) decrease in SpO2 of more than 10% below pre-procedure baseline during the 1-hour post-procedure.
  2. Persistent (>10 minute) increase in HR of more than 30 beats per minute above pre-procedure baseline during the 1-hour post-procedure.
  3. Persistent (>10 minute) decrease in MAP of more than 15 mm Hg below pre-procedure baseline during the 1-hour post-procedure.
Mean log transformed IL-10:IL-12p70 ratio in tracheal secretion, bronchial secretion, and serum between days 3-4 | Days 3 to 4 of mechanical ventilation
  Tracheal aspirates (TA), bronchial fluid (nb-BALF), and blood are collected within 48-hours following endotracheal intubation. All three samples are collected again at two additional time points following intubation: between days 3-4 and between days 5-7, so long as the patient remains endotracheally intubated. Three time points were chosen to show consistency in ratio of IL-10 to IL-12p70 between TA and nb-BALF throughout the first week of endotracheal intubation. If a patient is extubated before day 7 all sample collection will stop. No samples will be obtained after 7 days of intubation as we are focusing on the acute phase of lung injury only. An ELISA assay is performed to measure the concentration of IL-10 and IL-12p70 for ratio comparison.
Mean log transformed IL-10:IL-12p70 ratio in tracheal secretion, bronchial secretion, and serum between days 5-7 | Days 5 to 7 of mechanical ventilation
  Tracheal aspirates (TA), bronchial fluid (nb-BALF), and blood are collected within 48-hours following endotracheal intubation. All three samples are collected again at two additional time points following intubation: between days 3-4 and between days 5-7, so long as the patient remains endotracheally intubated. Three time points were chosen to show consistency in ratio of IL-10 to IL-12p70 between TA and nb-BALF throughout the first week of endotracheal intubation. If a patient is extubated before day 7 all sample collection will stop. No samples will be obtained after 7 days of intubation as we are focusing on the acute phase of lung injury only. An ELISA assay is performed to measure the concentration of IL-10 and IL-12p70 for ratio comparison.

OTHER OUTCOMES:
Fraction of screened patients enrolled, fraction of patients with complete sample collection, and fraction of patients with complete clinical data | 1-Year from Initial Enrollment
  Estimate the feasibility of enrolling ARDS patient for a future larger trial designed to examine IL-10:IL-12p70 as a predictor of ARDS in pediatric patients. This study will generate pilot data regarding consent rate, estimates of data completion, and fraction of missing clinical data necessary for us to determine whether a future study involving the ratio of IL-10 to IL-12p70 can be used as a predictor of ARDS in this population.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lercher, MD, Principal Investigator — University of North Carolina Hospital at Chapel Hill; Benny Joyner, MD, MPH, Study Director — University of North Carolina, Chapel Hill; Benny L Joyner, Jr., MD, MPH, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina, United States